CLINICAL TRIAL: NCT00808210
Title: A PHASE II RANDOMIZED, DOUBLE-BLIND, PARALLEL GROUP STUDY TO EVALUATE THE EFFICACY AND SAFETY OF OCRELIZUMAB IN COMBINATION WITH METHOTREXATE, COMPARED TO INFLIXIMAB PLUS METHOTREXATE IN PATIENTS WITH ACTIVE RHEUMATOID ARTHRITIS CURRENTLY RESPONDING INADEQUATELY TO ETANERCEPT OR ADALIMUMAB
Brief Title: A Study to Evaluate Ocrelizumab in Combination With Methotrexate Compared With Infliximab Plus Methotrexate in Patients With Active Rheumatoid Arthritis Currently Responding Inadequately to Etanercept or Adalimumab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on analysis of results and consideration of available treatments, the overall benefit to risk profile of ocrelizumab was not favorable in RA.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT4562g; GA00931
Record Dates: First submitted 2008-12-11; First posted 2008-12-15 (Estimated); Results first posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-10

CONDITIONS: Rheumatoid Arthritis
Keywords: RA; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Infliximab; Methotrexate; Methylprednisolone; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Ocrelizumab 200mg (Experimental): Participants received two intravenous (IV) infusions of 200 mg ocrelizumab administered on Day 1 and Day 15 and placebo IV infliximab infusions administered on Day 1, Day 15, Week 6, and Week 14. In addition to the study medication, all patients were to receive methotrexate at a stable dose of 7.5-25 mg/week and folic acid or equivalent at a dose of 5 mg/week to minimize methotrexate toxicity.
  Interventions: Drug: Methotrexate; Drug: Methylprednisolone; Drug: Ocrelizumab; Drug: Placebo
- Infliximab 5mg/kg (Active Comparator): Participants received four IV infusions of 5 mg/kg infliximab administered on Day 1, Day 15, Week 6, and Week 14 and placebo ocrelizumab infusions administered on Day 1 and Day 15. In addition to the study medication, all patients were to receive methotrexate at a stable dose of 7.5-25 mg/week and folic acid or equivalent at a dose of 5 mg/week to minimize methotrexate toxicity.
  Interventions: Drug: Infliximab; Drug: Methotrexate; Drug: Methylprednisolone; Drug: Placebo

INTERVENTIONS:
Drug: Infliximab — Intravenous repeating dose
  Arms: Infliximab 5mg/kg
Drug: Methotrexate — Oral or parenteral repeating dose
Drug: Methylprednisolone — Intravenous repeating dose
Drug: Ocrelizumab — Intravenous repeating dose
  Arms: Ocrelizumab 200mg
Drug: Placebo — Intravenous repeating dose

SUMMARY:
This is a Phase II, randomized, active-controlled, double-blind, double-dummy, parallel-group, multicenter study in the United States enrolling patients with active RA. The study will enroll approximately 290 patients at approximately 130 sites.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Current treatment for RA on an outpatient basis
* Active disease
* Currently receiving 50 mg etanercept subcutaneously (SC) every week or 40 mg adalimumab SC every other week.
* Considered by Investigator to be a primary non-responder to their first anti-TNFÎ± treatment for efficacy reasons

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA
* History of, or current, inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other systemic autoimmune disorder (e.g., systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease or other overlap syndrome)
* Previous treatment with a any biologic therapy for RA (including investigational products with the exception of etanercept or adalimumab
* Treatment with more than one prior anti-TNFÎ± therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-03-05 (Actual); Primary Completion 2012-11-14 (Actual); Study Completion 2012-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (53):
- United States (53):
  - Rheumatology Associates, Birmingham, Alabama
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Dr. Brigid Freyne, MD, Murrieta, California
  - Agilence Arthritis and Osteoporosis Medical Center, Inc., Whittier, California
  - Arthritis Assoc & Osteoporosis; Ctr of Colorado Springs, Colorado Springs, Colorado
  - RASF-Clinical Research Center, Boca Raton, Florida
  - Robert W. Levin MD - PP, Dunedin, Florida
  - Science and Research Institute, Inc., Jupiter, Florida
  - Rheumatology Associates of Central Florida, Orlando, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - Arthritis Res & Treatment, Macon, Georgia
  - Harbin Clinic, Rome, Georgia
  - Institute of Arthritis Research, Idaho Falls, Idaho
  - Illinois Bone & Joint Inst., Morton Grove, Illinois
  - Springfield Clinic, Springfield, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - Hurley Medical Center, Flint, Michigan
  - Rheumatology, P.C.; Medical Arts Building, Kalamazoo, Michigan
  - Fiechtner Research Inc, Lansing, Michigan
  - Shores Rheumatology, Saint Clair Shores, Michigan
  - Jackson Arthritis Clinic, Flowood, Mississippi
  - Arthritis Associates of Mississippi, Jackson, Mississippi
  - Private Practice - Rosenberg, Florissant, Missouri
  - Clayton Medical Research, St Louis, Missouri
  - Billings Clinic; Research Center, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Westroads Medical Group, Omaha, Nebraska
  - Arthritis Center of Reno, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Rheumatology 5C, Lebanon, New Hampshire
  - Regional Clinical Research, Binghamton, New York
  - Arthritis & Osteoporosis Center, Brooklyn, New York
  - Southern Tier Arthritis & Rheumatism, Olean, New York
  - Buffalo Rheumatology Associates, Orchard Park, New York
  - Barada,Harrell,Toohey&Bellhorn, Durham, North Carolina
  - Physicians East Pa, Greenville, North Carolina
  - Ohio State Univ Med Center, Columbus, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Healthcare Research Consultants, Tulsa, Oklahoma
  - Providence Arthritis Center, Portland, Oregon
  - Lehigh Valley Physicians Group, Allentown, Pennsylvania
  - Arthritis Associates, Erie, Pennsylvania
  - Columbia Arthritis Center (Partnership Practice), Columbia, South Carolina
  - Piedmont Arthritis Clinic, Greenville, South Carolina
  - South Carolina Research Center, Myrtle Beach, South Carolina
  - Arthritis Associates, Hixson, Tennessee
  - Ramesh Gupta - PP, Memphis, Tennessee
  - Ctr for Inflammatory Disease, Nashville, Tennessee
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Phillip A Waller MD, PA, Houston, Texas
  - Southwest Rheumatology, Mesquite, Texas
  - Texas Arthritis Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/members/ourmembers/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Period: Study Period + 48 Weeks of Follow-up
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Started | 15 | 13
Completed | 6 | 4
Not Completed | 9 | 9
Not completed — Sponsor decision to terminate study | 3 | 7
Not completed — Other reasons outside Sponsor decision | 6 | 2
Period: Double-Blind TX Period
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Started | 15 | 13
Completed | 13 | 10
Not Completed | 2 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Sponsor decision to terminate study | 1 | 1
Not completed — Other reasons outside Sponsor decision | 1 | 1
Period: Open Label Ocrelizumab Treatment Period
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Started | 9 | 4
Completed | 0 | 0
Not Completed | 9 | 4
Not completed — Sponsor decision to terminate study | 9 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (12.9) | 54.2 (15.2) | 53.83 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 9 | 3 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in DAS28(ESR) at Week 20
Time Frame: Week 20
Population: The study was terminated before data for the primary and secondary efficacy endpoints were collected so no data was collected for these efficacy endpoints.
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Participants With Clinical Response of 20% According to ACR Criteria
Time Frame: Baseline up to 30 months
Population: as for outcome 1
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With Clinical Response of 50% According to ACR Criteria
Time Frame: Baseline up to 30 months
Population: as for outcome 1
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Participants With Clinical Response of 70% According to ACR Criteria
Time Frame: Baseline up to 30 months
Population: as for outcome 1
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: European League Against Rheumatism (EULAR) Response Rates
Time Frame: Baseline up to 30 months
Population: as for outcome 1
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Time Frame: Baseline up to 30 months
Population: as for outcome 1
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Fatigue Visual Analog Scale Score (VAS)
Time Frame: Baseline up to 30 months
Population: as for outcome 1
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Time Frame: Baseline up to 30 months
Measure: Number; unit: Percentage of Participants
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
Number analyzed (Participants) | 15 | 13
Percentage of Participants | 78.9 | 76.9

ADVERSE EVENTS:
Time Frame: Baseline up to 43 months
Description: 4 patients from infliximab switched to ocrelizumab during the open label phase and the summary of AEs were summarized in the ocrelizumab arm for the safety analysis.
Arm/Group | Ocrelizumab 200mg | Infliximab 5mg/kg
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/13
Serious Adverse Events (participants affected / at risk) | 2/19 | 0/13
Other Adverse Events (participants affected / at risk) | 15/19 | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab 200mg (N=19) | Infliximab 5mg/kg (N=13)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HUMERUS FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.05% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab 200mg (N=19) | Infliximab 5mg/kg (N=13)
UPPER RESPIRATORY TRACT INFECTIOn (Infections and infestations) | 4 (4) | 1 (1)
SINUSITIS (Infections and infestations) | 3 (3) | 0 (0)
ALVEOLAR OSTEITIS (Infections and infestations) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0)
CYSTITIS (Infections and infestations) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 2 (2) | 0 (0)
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Infections and infestations) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0)
ORAL INFECTION (Infections and infestations) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 1 (1) | 0 (0)
TOOTH ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
ENTERITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 (1) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
COLD SWEAT (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ROSACEA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
CHILLS (General disorders) | 1 (1) | 2 (2)
FATIGUE (General disorders) | 0 (0) | 1 (1)
CHEST PAIN (General disorders) | 1 (1) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 0 (0) | 2 (2)
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 (0) | 1 (1)
HEAD TITUBATION (Nervous system disorders) | 0 (0) | 1 (1)
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1 (1) | 0 (0)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEART RATE INCREASED (Investigations) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
BENIGN NEOPLASM OF THYROID GLAND (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
TOOTH EXTRACTION (Surgical and medical procedures) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (1) | 0 (0)
JOINT DISLOCATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
At the time of study termination the scope of the statistical analyses was reduced and limited to evaluation of the safety profile.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights